CLINICAL TRIAL: NCT06550128
Title: Randomized, Multi-center Phase II Study to Evaluate the Efficacy and Safety of AHB-137 in HBeAg-negative CHB Subjects Under Stable Nucleos(t)Ide Analogue (NA) Treatment
Brief Title: Study to Evaluate the Efficacy and Safety of AHB-137 Injection in Participants With Chronic Hepatitis B (CHB).
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ausper Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB-10-8003
Record Dates: First submitted 2024-08-05; First posted 2024-08-12 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AHB-137 (Experimental)
  Interventions: Drug: AHB-137
- Placebo (Placebo Comparator)
  Interventions: Drug: AHB-137 and Placebo
- AHB-137 (16 weeks) (Experimental)
  Interventions: Drug: AHB-137 (16weeks)

INTERVENTIONS:
Drug: AHB-137 — AHB-137 injection will be administered subcutaneously.
  Arms: AHB-137
Drug: AHB-137 and Placebo — AHB-137and placebo will be administered subcutaneously.
  Arms: Placebo
Drug: AHB-137 (16weeks) — AHB-137 injection will be administered subcutaneously.
  Arms: AHB-137 (16 weeks)

SUMMARY:
AB-10-8003 is a randomized, multi-center phase II study to evaluate the efficacy and safety of AHB-137 in subjects with HBeAg-negative CHB under stable NA treatment.

DETAILED DESCRIPTION:
The study is to evaluate the efficacy and safety of AHB-137 in HBeAg-negative CHB subjects. The total duration of the study, including screening phase, treatment phase and follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

1. Participants voluntarily participate in the study, and sign the Informed Consent Form (ICF) prior to screening, able to complete the study and discontinue their NA therapy according to the protocol;
2. At least 18 years old at the time of signing of the informed consent;
3. Body Mass Index (BMI) between 18 to 32 kg/m^2(inclusive) ;
4. Participants who are Hepatitis B envelop antigen (HBeAg) negative during screening;
5. Participants whose serum HBsAg positive for at least 6 months prior to screening;
6. Participants who have stable on NA therapy at least 6 months prior to screening;
7. Participants with HBsAg concentration >100 IU/mL and≤3000 IU/mL, HBV DNA<100 IU/mL;
8. Participants with alanine aminotransferase (ALT)≤ 2x upper limit of normal (ULN);
9. For women of childbearing potential, she should be non-pregnant or non-lactating during screening, and participants (and partners) are willing to take effective contraceptive measures from the screening until the last visit or at least 6 months after the last dosing.

Exclusion Criteria:

1. Clinical significant abnormalities except Chronic HBV infection, such as acute coronary syndrome within 6 months before screening, evidence of major surgery, major or unstable heart disease, bleeding tendency or significant coagulation disorder within 3 months before screening;
2. Any clinically significant liver diseases, including but not limited to hepatitis caused by other pathogenic infections, hemochromatosis, Wilson disease, primary biliary cirrhosis, autoimmune liver diseases, alcoholic liver disease, severe non-alcoholic fatty liver disease, Drug-induced liver injury, etc.;
3. Participants with severe infection requiring intravenous anti-infection treatment 1 month before randomization;
4. Active hepatitis C, Human immunodeficiency virus (HIV) positive, syphilis positive;
5. Liver stiffness measurement (LSM) > 9.0 kPa when screening;
6. Diagnosed or suspected hepatocellular carcinoma;
7. The laboratory examination results are obviously abnormal;
8. History of vasculitis or signs and symptoms of potential vasculitis;
9. History of extrahepatic disease that may be related to HBV immune status;
10. Administration of immunosuppressants within 3 months prior to screening, except for short-term use (≤2 weeks) or topical/inhaled steroids. Administration of immunomodulators (thymosin) and cytotoxic drugs within 6 months prior to the first study intervention or have a history of vaccination within 1 month prior to screening or planned administration during the study.
11. Administration of any Interferon within 6 months prior to screening;
12. History of malignant tumor within the past 5 years;
13. Any suspicion of drug component allergy, or allergic constitution (various drug and food allergy, and judged by the investigator to be clinically significant) in participants;
14. Participants who have significant trauma or major surgery within 3 months before screening, or plan to perform surgery during the study;
15. Blood donation or blood loss more than 400 mL within 12 weeks before screening; Blood transfusion; Blood donation or blood loss not less than 200 mL within 1 month before screening;
16. Concurrently participating in another clinical study, or received an investigational product within the following time period prior to the first dosing day in the current study: 5 half-lives or twice the duration of the biological effect of the study treatment or 90 days;
17. Any oligonucleotide or siRNA treatments within 12 months prior to first dosing;
18. Any other circumstances or conditions for which the investigator considers that the participants are inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving HBsAg < limit of detection (LOD) 0.05 International Unit/mL (IU/mL) and HBV DNA < lower limit of quantitation (LLOQ) with or without anti-HBs seroconversion at the end of treatment. | Up to 24 weeks

SECONDARY OUTCOMES:
Proportion of participants achieving HBsAg lower than LOD and HBV DNA lower than LLOQ , regardless of whether HBsAg seroconversion is observed | At 8 weeks
Proportion of participants meeting NA treatment discontinuation criteria. | Up to 48 weeks
Changes of the score of hepatitis B quality of life instrument (HBQOL) compared with baseline | Up to 72 weeks
  This scale has 31 items, including 7 dimensions: psychological status, expected anxiety, vitality, shame, infectivity, health vulnerability, and viral response. Each item is scored on a 5-point scale, with higher scores indicating a more severe impact of hepatitis B on quality of life.
Percentage of participants with different levels of HBsAg reduction compared with baseline | Up to 72 weeks
Serum levels of HBV DNA, HBsAg, highly sensitive HBsAg, HBcrAg, HBV RNA, HBsAb, HBeAb and HBsAg-HBsAb. | Up to 72 weeks
The time from the discontinuation of NA treatment to virological relapse | Up to 72 weeks
The time from the discontinuation of NA treatment to clinical relapse | Up to 72 weeks
Sequencing of the Viral DNA and/or viral RNA analysis for detection of drug resistance of AHB-137 | Up to 24 weeks
Safety: number of participants with adverse events (TEAEs), serious adverse events (SAE) and clinically significant examination results, including laboratory examination, electrocardiogram (ECG) examination, physical examination and vital signs | Up to 72 weeks
Immunogenicity: number and percentage of participants with detectable anti-drug antibodies (ADA) | Up to 72 weeks
Changes of cytokine levels compared with baseline | Up to 72 weeks
The pharmacokinetic profile of AHB-137: Maximum concentration (Cmax) of AHB-137 in plasma | Up to 72 weeks
The pharmacokinetic profile of AHB-137: Area under the concentration-time curve (AUC) of AHB-137 | Up to 72 weeks
Plasma concentrations of AHB-137 | Up to 72 weeks
Proportion of participants maintaining sustained response. | Up to 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, Principal Investigator — The First Hospital of Jilin University; Jinlin Hou, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (6):
- China (6):
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - The third People's Hospital of Zhenjiang, Zhenjiang, Jiangsu
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - The First Hospital of Jilin University, Jilin

IPD SHARING:
Plan to Share IPD: No